CLINICAL TRIAL: NCT02281214
Title: Genome Analysis by Next Generation Sequencing in Personalisation of Lung Cancer Treatment
Brief Title: NGS Genome Analysis in Personalisation of Lung Cancer Treatment
Acronym: ALCAPONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-A01163-44
Record Dates: First submitted 2014-10-23; First posted 2014-11-03 (Estimated); Last update posted 2019-01-04 (Actual); Status verified 2018-12

CONDITIONS: Lung Cancer
Keywords: lung cancer, mutations; patients; mutations
MeSH Terms: conditions — Lung Neoplasms | interventions — Blood Specimen Collection; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- blood sample, biopsy (Experimental)
  Interventions: Other: blood sample, biopsy

INTERVENTIONS:
Other: blood sample, biopsy — Blood samples and tumor biopsies will taken from patients before treatment and when tumor progression on therapy for Next Generation Sequencing (NGS) mutation analysis

SUMMARY:
The identification of driver mutations in the epidermal growth factor receptor (EGFR) as the primary oncogenic event in a subset of lung adenocarcinomas led to a model of targeted treatment and genetic profiling of the disease. EGFR tyrosine kinase inhibitors (TKIs) confer remission in some patients, but use of the EGFR-TKIs is limited to patients with adenocarcinomas who have known activating EGFR mutations. And resistance to TKI treatment has become an increasingly important cause of treatment failure. Therefore, identification of the molecular components involved could lead to the development of effective therapy. Today only a limited number of genetic alterations are studied.

Next Generation Sequencing (NGS) has the potential of becoming an important tool in clinical and therapeutic decision-making in oncology owing to its enhanced sensitivity in DND mutation detection.

ELIGIBILITY:
Inclusion Criteria:

* patients of bronchial adénocarcinoma with metastases can benefit from first-line therapy - targeted therapy by tyrosine kinase inhibitor(TKI) for EGFR mutation and chemotherapy for non EGFR mutation)
* Patients with epidermoid cancer of the lungs can benefit from chemotherapy
* man and women
* age ≥ 18 years
* Patients have signed a written informed consent form
* Patients are affiliated to s social health insurance

Exclusion Criteria:

* Survival time ≤ 3 months
* Patients with cerebral metastases
* Patients could not benefit from treatment for others diseases
* Pregnancy or breast-feeding
* Incapacity to sign the consent form for psychiatric, behavioural disorders
* Private individuals of freedom or under tutelage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2014-10-24 (Actual); Primary Completion 2014-11-17 (Actual); Study Completion 2018-11-17 (Actual)

PRIMARY OUTCOMES:
search for EGFR, KRAS, BRAF, PIK3CA, HER2, ERBB2, AKT1... mutations and ALK, ROS rearrangements by NGS | search for EGFR, KRAS, BRAF, PIK3CA, HER2, ERBB2, AKT1,... mutations and ALK , ROS rearrangements by NGS methods before treatment and when tumor progression in patients with first line metastatic lung cancer therapy (chimiotherapy, targeted therapy)

SECONDARY OUTCOMES:
comparison of genome profiles (mutations and rearrangements) | comparison of genome profiles (EGFR, KRAS, BRAF, PIK3CA, HER2, ERBB2, AKT1, ...mutations and ALK , ROS rearrangements) between targeted therapy for EGFR mutation and chemotherapy for non EGFR mutation
  To compare gene profiles (EGFR, KRAS, BRAF, PIK3CA, HER2, ERBB2, AKT1, APC, ... mutations and ALK , ROS rearrangements) in primary lung tumors before treatment and when tumor progression on therapy according to treatment groups (targeted therapy for EGFR mutation and chemotherapy for non EGFR mutation) using NGS methods
tumor genetic profile (EGFR, KRAS, BRAF, PIK3CA, HER2, ERBB2, AKT1, APC, ... mutations and ALK , ROS rearrangements) and circulating DNA genetic profile (EGFR, KRAS, BRAF, PIK3CA, HER2, ERBB2, AKT1, APC, ... mutations and ALK , ROS rearrangements) | To compare tumor genetic profile (EGFR, KRAS, BRAF, PIK3CA, HER2, ERBB2, AKT1, APC, ... mutations and ALK , ROS rearrangements) with circulating DNA genetic profile (EGFR, KRAS, BRAF, PIK3CA, HER2, ERBB2, ...mutations and rearrangements using NGS methods

CONTACTS AND LOCATIONS:
Overall Officials: Bruno COUDERT, MD, PhD, Principal Investigator — Centre Georges François Leclerc
Locations (1):
- Centre Georges François Leclerc, Dijon, France

REFERENCES:
- [Derived] Dalens L, Niogret J, Richard C, Chevrier S, Foucher P, Coudert B, Lagrange A, Favier L, Westeel V, Kim S, Adotevi O, Chapusot C, Martin L, Arnould L, Kaderbhai CG, Boidot R. Durable response of lung carcinoma patients to EGFR tyrosine kinase inhibitors is determined by germline polymorphisms in some immune-related genes. Mol Cancer. 2023 Jul 29;22(1):120. doi: 10.1186/s12943-023-01829-4. PMID 37516818